CLINICAL TRIAL: NCT01796067
Title: Families Improving Together (FIT) for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: University of Michigan (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dawn Wilson, Professor, University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016136; R01HD072153 (NIH)
Record Dates: First submitted 2013-01-22; First posted 2013-02-21 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Overweight; Obese
Keywords: Motivational intervention; Positive Parenting Intervention; Obesity; Physical Activity; Diet; African American; Adolescent
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Mot. & Fam. Weight Loss + Online Interv. (Experimental): Participants are randomized to motivational and family weight loss program plus the online intervention.
  Interventions: Behavioral: Motivational and Family Weight Loss; Behavioral: Online Intervention
- Mot. & Fam. Weight Loss + Online Control (Experimental): Participants are randomized to motivational and family weight loss intervention and then the online control program.
  Interventions: Behavioral: Motivational and Family Weight Loss; Behavioral: Online Control
- Basic Health Educ. & Online Interv. (Experimental): Participants are randomized to the basic health education program and then the online intervention program.
  Interventions: Behavioral: Basic Health Education; Behavioral: Online Intervention
- Basic Health Educ. & Online Control (Active Comparator): Participants are randomized to the basic health education program and then to the online control program.
  Interventions: Behavioral: Basic Health Education; Behavioral: Online Control

INTERVENTIONS:
Behavioral: Motivational and Family Weight Loss — This group will receive the comprehensive motivational and family weight loss intervention.
  Arms: Mot. & Fam. Weight Loss + Online Control; Mot. & Fam. Weight Loss + Online Interv.
Behavioral: Basic Health Education — This group will receive the comprehensive basic health education intervention.
  Arms: Basic Health Educ. & Online Control; Basic Health Educ. & Online Interv.
Behavioral: Online Intervention — Participants will receive the online tailored weight loss intervention program after they have either received the motivational plus family weight loss program or basic health face-to-face program.
  Arms: Basic Health Educ. & Online Interv.; Mot. & Fam. Weight Loss + Online Interv.
Behavioral: Online Control — Participants will receive the online control program after they have either received the motivational plus family weight loss program or the basic health education program.
  Arms: Basic Health Educ. & Online Control; Mot. & Fam. Weight Loss + Online Control

SUMMARY:
The increasing rate of obesity has become a major public health concern with national reports indicating 40% of African American adolescents are now overweight/obese. Little is known about effective weight loss interventions in ethnic minority adolescents. However, research has shown that ethnic minorities attend fewer intervention sessions, have higher attrition rates and lose less weight compared to Caucasians. Two fundamental problems related to this lack of progress are 1) lack of appropriate content of weight loss interventions for African American adolescents that integrate cultural issues, parenting skills, and motivational strategies for long-term change and, 2) poor dose of weight loss interventions because of participant fatigue and drop out. While previous weight loss studies for adolescents have been long lasting (12-25 weeks), our team developed a weight loss program that is a relatively brief (8-week) face-to-face intervention that integrates motivational (autonomy-support) and positive parenting skills (monitoring, social support, positive communication skills) for reducing z-BMI in overweight African American adolescents. Our team recently conducted a pilot study testing the feasibility of an 8-week on-line culturally tailored intervention, Thus, the goal of this project is to conduct a randomized controlled efficacy trial to address the problems with past studies by 1) making the face-to-face group intervention shorter, 2) using an on-line component to compliment the group-based intervention for increasing dose, and by 3) tailoring a motivational and parenting skills program directly to parents and adolescents skill levels and cultural background. 520 overweight African American adolescents and their parents will be recruited to participate. Phase I of the trial will test the efficacy of an 8-week face-to-face group randomized trial comparing motivational plus family-based weight loss (M+FWL) to a basic health (BH) education program on reducing z-BMI and improving diet and physical activity (PA) in overweight African American adolescents. In phase II of the trial participants will be re-randomized to either an 8-week on-line intervention or a control on-line program resulting in a 2 (M+FWL vs. BH group) x 2 (intervention vs. control on-line program) factorial design. A 6-month follow-up will examine whether adolescents in the 8-week M+FWL group plus 8-week on-line intervention program will show the greatest maintenance in reducing z-BMI.

ELIGIBILITY:
Inclusion Criteria:

* Must have a parent or primary caregiver who lives in the same house as the adolescent
* Live within 60 miles of the program's office
* Have at least 3 grandparents who are African American
* Access to the internet
* Children between the ages of 11 and 16
* Child must have BMI above 85th percentile and below 99th percentile
* Have no medical condition that would limit participation in moderate intensity exercise including life-threatening illness (e.g., immobile, severely disabled, or bed ridden)
* Available and able to participate in measures and intervention activities over the next year

Exclusion Criteria:

* Adolescents with chronic illness
* Adolescents who require a specialized diet may not be eligible
* Developmental delay
* Partaking currently in another weight loss program

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2012-07; Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (z-BMI) in Adolescents | Baseline to 2 months
  We are investigating whether there is change in body mass index (BMI; age- and sex-adjusted based upon CDC norms) from baseline to 2 months and whether there are group differences (i.e., M+FWL vs. BH groups) in change in BMI in adolescents.
Change in Body Mass Index (z-BMI) in Adolescents | Baseline to 4 months
  We are investigating whether there is change in body mass index (BMI; age- and sex-adjusted based upon CDC norms) from baseline to 4 months and whether there are group differences (i.e., M+FWL & Intervention online, M+FWL & Control online, BH & Intervention online, BH & Control online) in change in BMI in adolescents.
Change in Body Mass Index (z-BMI) in Adolescents | Baseline to 6-month follow-up
  We are investigating intervention effects on change in body mass index (BMI; age- and sex-adjusted based upon CDC norms) from baseline to 6 months post-intervention. Specifically, we will examine whether there are group differences (i.e., M+FWL & Intervention online, M+FWL & Control online, BH & Intervention online, BH & Control online) in maintenance in BMI in adolescents.

SECONDARY OUTCOMES:
Change in Moderate to Vigorous Physical Activity (MVPA) in Parents and Adolescents | Baseline to 4 months
  Minutes per day; We are investigating whether there is change of physical activity from baseline to 4 months and whether there are group differences (i.e., M+FWL & Intervention online, M+FWL & Control online, BH & Intervention online, BH & Control online) in change in MVPA in parents and adolescents.
Change of 24 Hour Dietary Recall (NDRS) of Kcals in Parents and Adolescents | Baseline to 4 months
  We are investigating whether there is change of Kcals at 4 months. We are looking at these effects for fruit and vegetable intake, as well as total fat intake and whether there are group differences (i.e., M+FWL & Intervention online, M+FWL & Control online, BH & Intervention online, BH & Control online) in change in diet in parents and adolescents.
Change in Psychosocial Variables in Adolescents | Baseline to 4 months
  Examine the effects of psychosocial variables (autonomy-support, monitoring, communication) as potential mediators of the intervention effects on changes in z-BMI, dietary intake, and MVPA in adolescents.
Change in Moderate to Vigorous Physical Activity in Adolescents | Baseline to 6-month Follow-up
  Minutes per day; We are investigating whether there is change of physical activity at the 6-month follow-up and whether there are group differences (i.e., M+FWL & Intervention online, M+FWL & Control online, BH & Intervention online, BH & Control online) in change in MVPA in adolescents.
Change of 24 Hour Dietary Recall (NDRS) of Kcals in Adolescents | Baseline to 6-month Follow-up
  We are investigating whether there is change of Kcals at 6-month follow-up. We are specifically looking at effects for fruit and vegetable intake, as well as total fat intake in adolescents, and vegetable intake, as well as total fat intake and whether there are group differences (i.e., M+FWL & Intervention online, M+FWL & Control online, BH & Intervention online, BH & Control online) in change in diet in adolescents.
Change in Body Mass Index (z-BMI) in Parents | Baseline to 4 months
  We are investigating whether there is change in body mass index (BMI; age- and sex-adjusted based upon CDC norms) from baseline to 4 months and whether there are group differences (i.e., M+FWL & Intervention online, M+FWL & Control online, BH & Intervention online, BH & Control online) in change in BMI in parents.
Change in Body Mass Index (z-BMI) for Parents | Baseline to 6 Months Follow-up
  We are investigating whether there is change in body mass index (BMI; age- and sex-adjusted based upon CDC norms) from baseline to 6 months and whether there are group differences (i.e., M+FWL & Intervention online, M+FWL & Control online, BH & Intervention online, BH & Control online) in change in BMI in parents.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn K Wilson, PhD, Principal Investigator — University of South Carolina
Locations (1):
- Obesity Research Group, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Quattlebaum M, Sweeney AM, Wilson DK. Ecological predictors of family mealtime over time among overweight African American adolescent-parent dyads. J Behav Med. 2025 Aug;48(4):630-643. doi: 10.1007/s10865-025-00571-0. Epub 2025 May 15. PMID 40374860
- [Derived] Kipp C, Wilson DK, Brown A, Quattlebaum M, Loncar H, Sweeney AM, Abshire DA. Compounding effects of stress on diet, physical activity, and wellbeing among African American parents: a qualitative study to inform the LEADS health promotion trial. J Behav Med. 2024 Aug;47(4):647-661. doi: 10.1007/s10865-024-00477-3. Epub 2024 Mar 9. PMID 38460063
- [Derived] Sweeney AM, Wilson DK, Resnicow K, Van Horn ML, Kitzman H. Engagement With Tailored Physical Activity Content: Secondary Findings From the Families Improving Together for Weight Loss Randomized Controlled Trial. J Med Internet Res. 2023 Apr 12;25:e42581. doi: 10.2196/42581. PMID 37043271
- [Derived] Brown A, Wilson DK, Sweeney AM, van Horn ML, Zarrett N, Pate RR. Buffering effects of protective factors on light and moderate-to-vigorous physical activity among african american women. J Behav Med. 2023 Jun;46(3):405-416. doi: 10.1007/s10865-022-00360-z. Epub 2022 Oct 19. PMID 36260160
- [Derived] Loncar H, Wilson DK, Sweeney AM, Quattlebaum M, Zarrett N. Associations of parenting factors and weight related outcomes in African American adolescents with overweight and obesity. J Behav Med. 2021 Aug;44(4):541-550. doi: 10.1007/s10865-021-00208-y. Epub 2021 Mar 9. PMID 33751355
- [Derived] Kipp C, Wilson DK, Sweeney AM, Zarrett N, Van Horn ML. Effects of Parenting and Perceived Stress on BMI in African American Adolescents. J Pediatr Psychol. 2021 Aug 19;46(8):980-990. doi: 10.1093/jpepsy/jsab025. PMID 33738484
- [Derived] Brown A, Wilson DK, Sweeney AM, Van Horn ML. The Moderating Effects of Social Support and Stress on Physical Activity in African American Women. Ann Behav Med. 2021 Apr 7;55(4):376-382. doi: 10.1093/abm/kaaa051. PMID 32692356
- [Derived] Sweeney AM, Wilson DK, Loncar H, Brown A. Secondary benefits of the families improving together (FIT) for weight loss trial on cognitive and social factors in African American adolescents. Int J Behav Nutr Phys Act. 2019 May 24;16(1):47. doi: 10.1186/s12966-019-0806-5. PMID 31126345
- [Derived] Wilson DK, Sweeney AM, Law LH, Kitzman-Ulrich H, Resnicow K. Web-Based Program Exposure and Retention in the Families Improving Together for Weight Loss Trial. Ann Behav Med. 2019 Mar 20;53(4):399-404. doi: 10.1093/abm/kay047. PMID 30892641
- [Derived] Wilson DK, Kitzman-Ulrich H, Resnicow K, Van Horn ML, St George SM, Siceloff ER, Alia KA, McDaniel T, Heatley V, Huffman L, Coulon S, Prinz R. An overview of the Families Improving Together (FIT) for weight loss randomized controlled trial in African American families. Contemp Clin Trials. 2015 May;42:145-57. doi: 10.1016/j.cct.2015.03.009. Epub 2015 Mar 30. PMID 25835731